CLINICAL TRIAL: NCT02406625
Title: Clinical and Neural Changes Associated With Dialectical Behavioral Therapy in Adolescents With Suicidal Behaviors
Brief Title: Dialectical Behavioral Therapy in Adolescents With Suicidal Behaviors
Acronym: DBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Clinic per a la Recerca Biomédica (Other)
Collaborators: Santamarina Pérez, Pilar (Unknown); Romero Cela, María Soledad (Unknown); Méndez Blanco, Iria (Unknown); Font, Elena (Unknown)
Responsible Party: Principal Investigator, Marisol Picado Rossi, Ph.D., Fundacion Clinic per a la Recerca Biomédica
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DBT001
Record Dates: First submitted 2015-03-19; First posted 2015-04-02 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Suicidal Behaviors
MeSH Terms: interventions — Behavior Therapy

ARMS (3):
- Diaclectical Behavioral Therapy (Experimental): 15 adolescents with history of suicidal behaviors receiving Dialectical Behavioral Therapy.
  Interventions: Behavioral: Behavioral Therapy
- Support Therapy (Experimental): 15 adolescents with history of suicidal behaviors receiving Support Therapy.
  Interventions: Behavioral: Behavioral Therapy
- Controls (No Intervention): A group of 15 healthy controls that are not receiving any kind of therapy.

INTERVENTIONS:
Behavioral: Behavioral Therapy — 16 therapeutic group sessions are delivered to both parents and adolescents; according to the assigned group for each family.
  Arms: Diaclectical Behavioral Therapy; Support Therapy

SUMMARY:
Suicidal behaviors among adolescents represents a public health problem due to its high prevalence and its low predictability. It is also known that brain development continues during adolescence, therefore, a therapeutic intervention during this period might propitiate neural changes that might favor the emotional regulation involved in suicidal behaviors. Dialectical Behavioral Therapy has proved to be effective regarding this problem.

For this reason, the investigators aimed to study the clinical, neuropsychological and neural effects of Dialectical Behavioral Therapy in adolescents with suicidal behaviors.

DETAILED DESCRIPTION:
Suicidal behaviors represent a public health problem due to its high prevalence and its low predictability. At a neurological level, higher vulnerability for suicidal behavior has been related to a frontostriatal-cingulum tract dysfunction as well as attention, memory and executive deficits. It is also known that brain development continues during adolescence, therefore, a therapeutic intervention during this period might propitiate neural changes that could favor the emotional regulation involved in suicidal behaviors. Specifically, Dialectical Behavioral Therapy has proved to be effective regarding this problem.

The investigators hypothesis is that DBT (Dialectical Behavioral Therapy) will improve clinical symptoms associated with suicidal behaviors, as well as the neural interconnections, which will result not only in structural and functional connectivity changes, but also in a better cognitive functioning. The investigators aimed to investigate the clinical, neuropsychological, and neural effects of Dialectical Behavioral Therapy in adolescents with suicidal behaviors.

The investigators method is a randomized, controlled study that includes 30 patients with suicidal behaviors and 15 healthy controls between the ages of 12 and 18 years. Patients were assigned to one of two groups (randomized): DBT and Regular Support Therapy. Clinical and neuropsychological evaluations were performed before and after the treatment for both patient groups. Additionally, Structural MRI data sets, diffusion-tensor imaging (DTI) and Functional Connectivity (Resting State fmri) were acquired for all patients and controls at baseline and after treatment. Initial characteristics will be compared between the three groups, and the investigators will also compared clinical, neuropsychological and imaging measures before and after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age between 12 and 18 years,
* Intellectual level over 70 (IQ>70)
* For the experimental groups:

  * Patients with suicidal behavior:

    * Real attempt,
    * Interrupted attempt,
    * Aborted attempt or behaviors, or
    * Preparation actions (based on the Columbia Suicide Severity Rating Scale -C-SSRS criteria) present during the last 12 months and that persist in the actual moment.

Exclusion Criteria:

* Presence of Acute Psychosis,
* Eating Disorder with an BMI < 18.5;
* Substance abuse in the current moment or during the last 6 months;
* Any neurological condition that curses with cognitive alterations; and
* Pregnancy.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 52 (Estimated)
Dates: Start 2014-11; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Clinical changes after 16 sessions of Dialectical Behavioral Therapy. | 4 months
  Clinical evaluations will be performed before and after the treatment in order to determine clinical improvement in relation to the applied therapy.
Neural changes after 16 sessions of Dialectical Behavioral Therapy. | 4 months
  Magnetic Resonance Imaging and functional Magnetic Resonance Imaging data sets will be acquired at baseline and then after the treatment, in order to determine anatomical or functional brain connectivity changes in relation to the applied therapy.
Neuropsychological changes after 16 sessions of Dialectical Behavioral Therapy. | 4 months
  Neuropsychological evaluations will be administrated before and after the treatment in order to determine changes in memory, attention or executive functioning in relation to the applied therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínic, Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Interventions for self-harm in children and adolescents. Cochrane Database Syst Rev. 2021 Mar 7;3(3):CD013667. doi: 10.1002/14651858.CD013667.pub2. PMID 33677832
- [Derived] Santamarina-Perez P, Mendez I, Singh MK, Berk M, Picado M, Font E, Moreno E, Martinez E, Morer A, Borras R, Cosi A, Romero S. Adapted Dialectical Behavior Therapy for Adolescents with a High Risk of Suicide in a Community Clinic: A Pragmatic Randomized Controlled Trial. Suicide Life Threat Behav. 2020 Jun;50(3):652-667. doi: 10.1111/sltb.12612. Epub 2020 Jan 16. PMID 31944371